CLINICAL TRIAL: NCT05499871
Title: Comparison Between Gait Retraining Intervention With a Transitioning Toward Minimalist Footwear on the Foot-ankle Strength, Running Economy and Injury Incidence in Endurance Runners: a One-year Follow up Study.
Brief Title: Effect of a Gait Retraining Intervention and a Minimalist Footwear Transition on Foot-ankle Strength, Running Economy and Injury in Endurance Runners.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Abran Guillaume, PhD student, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09082022
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Running; Wounds and Injuries; Oxygen Consumption
Keywords: Gait retraining; Performance; Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Minimalist footwear (Experimental): Transition toward a minimalist footwear.
  Interventions: Device: Transition to minimalist footwear.
- Footstrike pattern (Experimental): Transition toward a forefootstrike pattern.
  Interventions: Behavioral: Gait retraining intervention
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Gait retraining intervention — Participants will receive a training to modify their footstrike pattern toward a more forefoot strike and increase their cadence by 7.5%.
  Arms: Footstrike pattern
Device: Transition to minimalist footwear. — Participants will receive a running minimalist footwear.
  Arms: Minimalist footwear

SUMMARY:
The main aim is to determine whether a gait retraining intervention will improve the strength of the foot-ankle muscle, the running economy and reduce the injury incidence in a one-year follow-up study. The secondary aim is to seek whether a minimal foot-ankle strength is necessary to reduce the risk to sustain to a running-related-injury to transit toward a forefoot strike pattern or toward a minimalist footwear for an endurance runner.

Participants will be assessed at baseline, at 2 month follow-up, at 6 month follow-up and at 12 month follow-up. Assessment will be composed by questionnaires, a foot screening, maximal voluntary isometric strength of foot-ankle muscle with hand held dynamometer. Then, participants will run on a treadmill at self-paced and at 10 km/h with to measure their running economy and their footstrike pattern. In function of their distribution, participants will receive either nothing (control group) or minimalist footwear or a training to modify their footstrike pattern toward a more forefoot strike.

ELIGIBILITY:
Inclusion Criteria:

* Run 15 km per week since minimum 6 month

Exclusion Criteria:

* No running related injuries in the last 3 month before the participation.
* Have never worn minimalist footwear (minimalist index superior to 70%)
* Have never modified their footstrike pattern

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in foot-ankle strength | Change from Baseline foot-ankle strength at 2 month follow-up, Change from Baseline foot-ankle strength at 6 month follow-up, Change from Baseline foot-ankle strength at 12 month follow-up
  Measure of maximal voluntary isometric strength of ankle plantar flexors, hallux flexors, lesser toe flexors with hand held dynamometer.
Change in running economy | Change from Baseline running-economy at 2 month follow-up, Change from Baseline running economy at 6 month follow-up, Change from Baseline running economy at 12 month follow-up
  Measure of oxygen uptake was during steady state run on a treadmill at 10 km/h and at self-paced with was recorded using Ergocard device. Then, running economy was caluled with the formula: Energetic cost = 16.89 * Vo2 + 4.84*VCo2
Running-related-injuries | At any time during the 12 month follow-up
  Number of running related injuries per participant

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume Abran, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abran G, Schwartz C, Dardenne N, Delvaux F, Croisier JL. Minimalist Footwear and Softer Running Technique Alter Injury Location but Not Incidence in Recreational Endurance Runners. Am J Sports Med. 2026 Jan;54(1):109-117. doi: 10.1177/03635465251392242. Epub 2026 Jan 1. PMID 41476413